CLINICAL TRIAL: NCT05469022
Title: A Phase II, Single-Center, Single-Arm, Prospective Study of Neoadjuvant Lazertinib Therapy in Resectable EGFR-Mutation Positive Lung Adenocarcinoma Patients Detected by Broncho-alveolar Lavage Fluid(BALF) Liquid Biopsy
Brief Title: Neoadjuvant Lazertinib Therapy in EGFR-Mutation Positive Lung Adenocarcinoma Detected by BALF Liquid Biopsy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Collaborators: Yuhan Corporation (Industry)
Responsible Party: Principal Investigator, Kye Young Lee, Professor, Konkuk University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeolazBAL
Record Dates: First submitted 2022-07-15; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR mutation; extracellular vesicle; bronchoalveolar lavage; liquid biopsy; lazertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Lazertinib (Experimental): Lazertinib as neoadjuvant treatment is administrated for 9 weeks before surgery. After surgical intervention the treatment is administrated upto 3 years to the patients with over stage 2 tumor. Treatment is discontinued in case of unacceptable toxicity or disease progression.
  Interventions: Drug: Neoadjuvant lazertinib

INTERVENTIONS:
Drug: Neoadjuvant lazertinib — Lazertinib 240mg p.o once daily.
  Other Names: Neoadjuvant LECLAZA

SUMMARY:
Complete surgical resection is the standard treatment in early-stage lung cancer. However, the patients with early resected Epidermal Growth Factor Receptor(EGFR)-mutated lung cancers have high recurrence rate. The efficacy of neoadjuvant treatment by first-generation EGFR-Tyrosine Kinase Inhibitor(TKI) has been demonstrated, however, that of the third-generation EGFR-TKI(lazertinib) has not yet been fully investigated. The aim of this study is to evaluate the efficacy of neoadjuvant Lazertinib in resectable EGFR mutation-positive NSCLC and clinical application of extracellular vesicles(EVs) based BALF liquid biopsy to identify EGFR mutation without invasive tissue biopsy.

DETAILED DESCRIPTION:
The neoadjuvant treatment of 3rd-generation EGFR-TKI, lazertinib for 9 weeks before surgery is administrated. After the surgery, the patients with the tumor over stage 2 are given the lazertinib to prevent recurrence for 3 years or until recurrence. In early lung cancer, a tissue biopsy is often difficult due to the small size or the risky location. We collect bronchoalveolar lavage fluid for liquid biopsy and lazertinib is administrated according to the result of BALF liquid EGFR genotyping.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years
2. Patients with suspected lung cancer on chest CT findings
3. Patients with the following EGFR gene mutations in the test on bronchoalveolar lavage fluid: E19Del, L858R alone or concurrent rare EGFR gene mutations (T790M, G719X, exon 20 insertion, S768I)
4. Patients whose tumor can be completely resected by surgery: patients with stage I-IIIB, or stage IVA who has single metastasis
5. Patients not previously treated with EGFR-TKIs such as gefitinib, erlotinib, afatinib, dacomitinib
6. Patients with the measurable lesion of 1 cm or more according to RECIST v1.1
7. Eastern Cooperative Oncology Group (ECOG) 0-1
8. EGFR-TKIs (gefitinib, erlotinib, afatinib,dacomitinib) naive patients
9. Patients with adequate pulmonary and heart function for surgery
10. Adequate organ function defined as Hemoglobin ≥ 9.0g/dL Absolute neutrophil count ≥ 1500/mm3 Platelet ≥ 100,000 /mm3 Serum creatinine≤ normal range*1.5x Aminotransferase/Alkaline phosphatase ≤normal range*2.5x Total bilirubin ≤1.5 mg/dL Liver metastasis: Aminotransferase/Alkaline phosphatase ≤ normal range* 5x Bone metastasis Alkaline phosphatase ≤ normal range* 5x
11. Female patients with childbearing potential should be using adequate contraceptive measures. Female patients must have evidence of non-child-bearing potential(Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments)
12. Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception for at least 14 days prior to administration of the first dose of study treatment, during the study, and for 3 months following the last dose of Lazertinib.

Exclusion Criteria:

1. Uncontrolled active interstitial lung disease
2. Pathologically confirmed N3 disease
3. Uncontrolled stage III-IV other malignancy
4. Uncontrolled Hypertension, Congestive Heart failure with New York Heart Association(NYHA) ≥ 3, acute myocardial infarct history within 6 months before screening. 2nd- 3rd Atrio-Ventricular(AV) block or complete AV block
5. Gastrointestinal diseases (e.g. Chron's disease, ulcerative colitis) or malabsorption syndrome that would impact on drug absorption
6. Active infection requiring ongoing treatment(e.g. active Hepatitis B virus, Hepatitis C virus or Human immunodeficiency virus)
7. History of hypersensitivity to active or inactive excipients of Lazertinib or drugs with a similar chemical structure.
8. No ability to comply with protocol requirements.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-05-19 (Estimated); Study Completion 2027-05-19 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 9 weeks after the starting day of the lazertinib
  The objective response rate (ORR) evaluated with RECIST version 1.1. It is defined as the proportion of patients with complete response (CR) or partial response (PR) after 9 weeks of lazertinib administration

SECONDARY OUTCOMES:
Down-staging rate | From the day of screening to an average of 16 weeks after the first dose
  The rate of downstage by pathology stage compared with clinical stage
Major pathological response | From the day of screening to an average of 16 weeks after the first dose
  The proportion of patients with less than 10% of the cancer cells in the surgical sample.
Disease-free survival rate | up to 3 years after surgery
  The length of time after surgical resection the patient remains free of recurrence/progression or death, whatever the cause.
The concordance rate of EGFR mutations between surgical tissue and BAL fluid samples | From the day of screening day to an average of 16 weeks after the first dose
  The concordance rate of BALF EGFR mutation compared with EGFR mutation status of surgical resected tissue

CONTACTS AND LOCATIONS:
Overall Officials: Kye Young Lee, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Zhong WZ, Wang Q, Mao WM, Xu ST, Wu L, Shen Y, Liu YY, Chen C, Cheng Y, Xu L, Wang J, Fei K, Li XF, Li J, Huang C, Liu ZD, Xu S, Chen KN, Xu SD, Liu LX, Yu P, Wang BH, Ma HT, Yan HH, Yang XN, Zhou Q, Wu YL; ADJUVANT investigators. Gefitinib versus vinorelbine plus cisplatin as adjuvant treatment for stage II-IIIA (N1-N2) EGFR-mutant NSCLC (ADJUVANT/CTONG1104): a randomised, open-label, phase 3 study. Lancet Oncol. 2018 Jan;19(1):139-148. doi: 10.1016/S1470-2045(17)30729-5. Epub 2017 Nov 21. PMID 29174310
- [Background] Xie H, Wang H, Xu L, Li M, Peng Y, Cai X, Feng Z, Ren W, Peng Z. Gefitinib Versus Adjuvant Chemotherapy in Patients With Stage II-IIIA Non-Small-Cell Lung Cancer Harboring Positive EGFR Mutations: A Single-Center Retrospective Study. Clin Lung Cancer. 2018 Nov;19(6):484-492. doi: 10.1016/j.cllc.2018.05.007. Epub 2018 May 26. PMID 30369426
- [Background] Yue D, Xu S, Wang Q, Li X, Shen Y, Zhao H, Chen C, Mao W, Liu W, Liu J, Zhang L, Ma H, Li Q, Yang Y, Liu Y, Chen H, Wang C. Erlotinib versus vinorelbine plus cisplatin as adjuvant therapy in Chinese patients with stage IIIA EGFR mutation-positive non-small-cell lung cancer (EVAN): a randomised, open-label, phase 2 trial. Lancet Respir Med. 2018 Nov;6(11):863-873. doi: 10.1016/S2213-2600(18)30277-7. Epub 2018 Aug 24. PMID 30150014
- [Background] Liu SY, Zhang JT, Zeng KH, Wu YL. Perioperative targeted therapy for oncogene-driven NSCLC. Lung Cancer. 2022 Oct;172:160-169. doi: 10.1016/j.lungcan.2022.05.007. Epub 2022 May 21. PMID 35644704
- [Background] Pennell NA, Neal JW, Chaft JE, Azzoli CG, Janne PA, Govindan R, Evans TL, Costa DB, Wakelee HA, Heist RS, Shapiro MA, Muzikansky A, Murthy S, Lanuti M, Rusch VW, Kris MG, Sequist LV. SELECT: A Phase II Trial of Adjuvant Erlotinib in Patients With Resected Epidermal Growth Factor Receptor-Mutant Non-Small-Cell Lung Cancer. J Clin Oncol. 2019 Jan 10;37(2):97-104. doi: 10.1200/JCO.18.00131. Epub 2018 Nov 16. PMID 30444685
- [Background] Zhang Y, Fu F, Hu H, Wang S, Li Y, Hu H, Chen H. Gefitinib as neoadjuvant therapy for resectable stage II-IIIA non-small cell lung cancer: A phase II study. J Thorac Cardiovasc Surg. 2021 Feb;161(2):434-442.e2. doi: 10.1016/j.jtcvs.2020.02.131. Epub 2020 Mar 19. PMID 32340810
- [Background] Xiong L, Li R, Sun J, Lou Y, Zhang W, Bai H, Wang H, Shen J, Jing B, Shi C, Zhong H, Gu A, Jiang L, Shi J, Fang W, Zhao H, Zhang J, Wang J, Ye J, Han B. Erlotinib as Neoadjuvant Therapy in Stage IIIA (N2) EGFR Mutation-Positive Non-Small Cell Lung Cancer: A Prospective, Single-Arm, Phase II Study. Oncologist. 2019 Feb;24(2):157-e64. doi: 10.1634/theoncologist.2018-0120. Epub 2018 Aug 29. PMID 30158288
- [Background] Zhong W, Yang X, Yan H, Zhang X, Su J, Chen Z, Liao R, Nie Q, Dong S, Zhou Q, Yang J, Tu H, Wu YL. Phase II study of biomarker-guided neoadjuvant treatment strategy for IIIA-N2 non-small cell lung cancer based on epidermal growth factor receptor mutation status. J Hematol Oncol. 2015 May 17;8:54. doi: 10.1186/s13045-015-0151-3. PMID 25981169
- [Background] Zhong WZ, Chen KN, Chen C, Gu CD, Wang J, Yang XN, Mao WM, Wang Q, Qiao GB, Cheng Y, Xu L, Wang CL, Chen MW, Kang X, Yan W, Yan HH, Liao RQ, Yang JJ, Zhang XC, Zhou Q, Wu YL. Erlotinib Versus Gemcitabine Plus Cisplatin as Neoadjuvant Treatment of Stage IIIA-N2 EGFR-Mutant Non-Small-Cell Lung Cancer (EMERGING-CTONG 1103): A Randomized Phase II Study. J Clin Oncol. 2019 Sep 1;37(25):2235-2245. doi: 10.1200/JCO.19.00075. Epub 2019 Jun 13. PMID 31194613
- [Background] Ahn MJ, Han JY, Lee KH, Kim SW, Kim DW, Lee YG, Cho EK, Kim JH, Lee GW, Lee JS, Min YJ, Kim JS, Lee SS, Kim HR, Hong MH, Ahn JS, Sun JM, Kim HT, Lee DH, Kim S, Cho BC. Lazertinib in patients with EGFR mutation-positive advanced non-small-cell lung cancer: results from the dose escalation and dose expansion parts of a first-in-human, open-label, multicentre, phase 1-2 study. Lancet Oncol. 2019 Dec;20(12):1681-1690. doi: 10.1016/S1470-2045(19)30504-2. Epub 2019 Oct 3. PMID 31587882
- [Background] Schaake EE, Kappers I, Codrington HE, Valdes Olmos RA, Teertstra HJ, van Pel R, Burgers JA, van Tinteren H, Klomp HM. Tumor response and toxicity of neoadjuvant erlotinib in patients with early-stage non-small-cell lung cancer. J Clin Oncol. 2012 Aug 1;30(22):2731-8. doi: 10.1200/JCO.2011.39.4882. Epub 2012 Jul 2. PMID 22753915
- [Background] Kim IA, Hur JY, Kim HJ, Kim WS, Lee KY. Extracellular Vesicle-Based Bronchoalveolar Lavage Fluid Liquid Biopsy for EGFR Mutation Testing in Advanced Non-Squamous NSCLC. Cancers (Basel). 2022 May 31;14(11):2744. doi: 10.3390/cancers14112744. PMID 35681723
- [Background] Kim IA, Hur JY, Kim HJ, Lee SE, Kim WS, Lee KY. Liquid biopsy using extracellular vesicle-derived DNA in lung adenocarcinoma. J Pathol Transl Med. 2020 Nov;54(6):453-461. doi: 10.4132/jptm.2020.08.13. Epub 2020 Oct 8. PMID 33027851
- [Background] Hur JY, Lee JS, Kim IA, Kim HJ, Kim WS, Lee KY. Extracellular vesicle-based EGFR genotyping in bronchoalveolar lavage fluid from treatment-naive non-small cell lung cancer patients. Transl Lung Cancer Res. 2019 Dec;8(6):1051-1060. doi: 10.21037/tlcr.2019.12.16. PMID 32010582